CLINICAL TRIAL: NCT04688086
Title: A Prospective Study to Evaluate the Effectiveness of Thermalytix (AI-based Thermographic Solution Developed by Niramai) for Breast Cancer Screening as Compared to Standard Screening Modalities for Breast Cancer
Brief Title: A Prospective Study to Evaluate Clinical Performance of Thermalytix in Detecting Breast Cancers
Status: Completed | Type: Observational
Sponsor: Niramai Health Analytix Private Limited (Industry)
Collaborators: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: NIR-THERMA-02
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Early Detection of Cancer
Keywords: Breast cancer; Thermography; Thermalytix; Artificial Intelligence; Machine Learning; Dense Breasts; Breast Density; Mammography; Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with no personal history of breast cancer: Women who came in for a breast mammography between ages 30 and 80 years were invited to take part in the study. All the women included in the study underwent breast cancer screening first by Thermalytix, the AI-based thermal imaging test, followed by mammography.
  Interventions: Diagnostic Test: Thermalytix

INTERVENTIONS:
Diagnostic Test: Thermalytix — Thermalytix is an Artificial intelligence based automated breast screening solution that analyzes thermal distribution on the breast to generate a breast health score automatically. Thermal imaging was performed by a trained technician to capture thermal images of the participant in five views. These thermal images were uploaded to Thermalytix software on the cloud where it was automatically analyzed by AI-based Thermalytix computer-aided detection (CADe) engine. This CADe engine analyzes uploaded thermal images and outputs an interpretation report for each participant with quantitative scores corresponding to computed probability of malignancy based on the structural, vascular, areolar, thermal properties of the observed abnormality. Thermalytix also generates annotated images with markings of abnormal regions and an overall Thermalytix score suggesting likelihood of breast malignancy. The locked AI model Thermalytix algorithm version 3, dated December 2018 was used for the analysis.

SUMMARY:
The purpose of this study is to determine the clinical performance of AI-based Thermalytix with the current standard-of-care diagnostic modalities in women.

DETAILED DESCRIPTION:
While mammography is the most accepted breast cancer screening test, it is less sensitive in women with dense breast tissue, who have a four fold high risk for developing breast cancer. Thermalytix is a novel automated breast cancer screening solution that uses artificial intelligence (AI) over thermal images to detect and localise breast cancer lesions in women. In this study the performance of Thermalytix over mammography is evaluated in women with dense and non-dense breast tissue who presented for a health check-up at a hospital. All women underwent Thermalytix and mammography, and participants who were reported as positive on either test were recommended for further investigations. Sensitivity, specificity, positive predictive value, and negative predictive value were calculated across age-groups, menopausal status, and breast densities against the current standard-of-care diagnostic modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects equal to and above 18 years
2. Subjects who are willing to give written informed consent for study participation
3. Subjects who are ready to comply with the study related visits and procedures

Exclusion Criteria:

1. Subjects who are pregnant
2. Subjects who are lactating
3. Subjects who have undergone either lumpectomy or mastectomy
4. Subjects who have undergone chemotherapy in the last 2 weeks at the time of study enrollment
5. Any active illness, psychological and/or pathological condition that would interfere with study participation in the opinion of the Investigator

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant eligibility is based on self-representation of gender identity
Study Population: Women who came in for a breast mammography at Max Super Speciality Hospital, Saket were invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richa Bansal, MD, Principal Investigator — Max Healthcare Insititute Limited
Locations (1):
- Max Healthcare Insititute Limited, New Delhi, India

IPD SHARING:
Plan to Share IPD: No
The study protocol and clinical study report will be made available to investigators from academic institutions for non-commercial use and whose proposed use of the data has been approved by an independent review committee. The individual participant data would be shared for meta-analysis.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With no Personal History of Breast Cancer
Started | 687
Completed | 459
Not Completed | 228
Not completed — Lost to Follow-up | 164
Not completed — Imaging error; | 64

BASELINE CHARACTERISTICS:
Population: Women with no personal history of breast cancer
Arm/Group | Women With no Personal History of Breast Cancer
Number analyzed (Participants) | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 441
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 459
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 459

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value of Thermalytix
Description: To assess the clinical performance of Thermalytix as compared to standard screening modalities.
  Sensitivity, specificity, positive predictive value and negative predictive value of Thermalytix
Time Frame: 2 days
Population: All women who satisfied the inclusion criteria
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Women With no Personal History of Breast Cancer
Number analyzed (Participants) | 459
percentage
  Sensitivity | 95.24 [76.18 to 99.88]
  Specificity | 88.58 [85.23 to 91.41]
  PPV | 28.57 [18.4 to 40.62]
  NPV | 99.74 [98.58 to 99.99]

2. Secondary Outcome: Sensitivity and Specificity of Thermalytix for Women With Dense Breast Tissue (ACR Category C or D)
Description: To assess the influence of patient characteristics (Breast density) on the diagnostic accuracy of Thermalytix.
Time Frame: 2 days
Population: Women with breast density ACR category C or D
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Women With no Personal History of Breast Cancer
Number analyzed (Participants) | 168
percentage
  Sensitivity | 100 [69.15 to 100]
  Specificity | 81.65 [74.72 to 87.35]

3. Secondary Outcome: Sensitivity and Specificity of Thermalytix in Women With Breast Density ACR Category "A" or "B"
Description: To assess the influence of patient characteristics (Breast density) on the diagnostic accuracy of Thermalytix.
  Sensitivity and Specificity of Thermalytix in Women with Fatty Breasts - Breast Density ACR category "A" or "B"
Time Frame: 2 days
Population: Women with Breast Density ACR category "A" or "B"
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Women With no Personal History of Breast Cancer
Number analyzed (Participants) | 291
percentage
  Sensitivity | 90.9 [73.9 to 100]
  Specificity | 92.5 [89.4 to 95.6]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of one year post study. No adverse events were reported during this period Each participant would require less than a day to assess if there was an adverse event.
Description: Self reported events.
Arm/Group | Women With no Personal History of Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/459
Serious Adverse Events (participants affected / at risk) | 0/459
Other Adverse Events (participants affected / at risk) | 0/459

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04688086/Prot_SAP_000.pdf